CLINICAL TRIAL: NCT06794294
Title: A Single Center, Open Label, Phase 1/2a Study to Evaluate Safety and Exploratory Efficacy of Allogenic Umbilical Cord Derived Mesenchymal Stem Cell Treatment in Patients with Rotator Cuff Disease
Brief Title: Effects of Allogenic Umbilical Cord-Derived Mesenchymal Stem Cells on Patients with Rotator Cuff Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASB-IP-001
Record Dates: First submitted 2025-01-13; First posted 2025-01-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients diagnosed with partial-thickness rotator cuff tear (Experimental)
  Interventions: Biological: Injection allogenic Umbilical Cord-derived Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Injection allogenic Umbilical Cord-derived Mesenchymal Stem Cell — Biological: Allogenic Umbilical Cord - derived Mesenchymal Stem Cell
  1. Injection dosage and volume of the study drugs:
     * Low dose: 1x10⁷ cells/3mL
  2. Number of injections: Only once during the study period
  3. Device: Ultrasound
  4. Injection technique: Injection into the lesion by investigator
  Biological: Allogenic Umbilical Cord - derived Mesenchymal Stem Cell
  1. Injection dosage and volume of the study drugs:
     * Mid dose: 5x10⁷ cells/3mL
  2. Number of injections: Only once during the study period
  3. Device: Ultrasound
  4. Injection technique: Injection into the lesion by investigator
  Biological: Allogenic Umbilical Cord - derived Mesenchymal Stem Cell
  1. Injection dosage and volume of the study drugs:
     * High dose: 1x10e8 cells/3mL
  2. Number of injections: Only once during the study period
  3. Device: Ultrasound
  4. Injection technique: Injection into the lesion by investigator

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Allogenic Umbilical Cord-derived Mesenchymal Stem Cell in Patients with Rotator Cuff Disease

ELIGIBILITY:
Inclusion Criteria:

* Male or female 19 years of age and older.
* Patients with unilateral shoulder pain lasting for at least 3months
* Patients who do not respond to conservative treatment.
* Patients who have not responded to sufficient non-surgical treatments, including medication, injection therapy, physical therapy, or exercise therapy, for more than 3 months
* Patients who have a partial-thickness rotator cuff tear confirmed with magnetic resonance imaging (MRI) or ultrasonography (US).
* Patients without any restrictions on clinical trial procedures, including hospitalization.

Exclusion Criteria:

* Patients who have received subacromial injection therapy on the affected shoulder within the past 3 months.
* Patients who have undergone rotator cuff surgery on the affected shoulder within the past 6 months
* Patients with a history of receiving stem cell therapy for the shoulder.
* Patients with the following shoulder conditions: complete rotator cuff tear, adhesive capsulitis, or isolated acromioclavicular joint arthropathy.
* Patients showing or suspected of having the following radiological findings: malignancy, severe osteoarthritis of the glenohumeral joint, or skeletal abnormalities decreasing the subacromial space.
* Patients presenting with symptomatic cervical spine disorders.
* Patients with concurrent bilateral shoulder pain
* Patients with polyarthritis, infectious arthritis, rheumatoid arthritis, or fibromyalgia.
* Patients with neurological deficit
* Pregnant women or lactating mothers.
* Patients unwilling to use effective contraception during the clinical trial period.
* Patients with current HBV, HCV, or HIV infections, or those with a positive RPR test.
* Patients with severe diseases that may affect the clinical trial, including cardiovascular disease, renal disease, liver disease, endocrine disorders, or malignancies.
* Patients who are unable to understand the questionnaires used for assessing their clinical status, including the Visual Analogue Scale (VAS), or those with psychiatric disorders impairing communication.
* Patients who do not wish to participate in the clinical trial or are unable to comply with follow-up schedules.
* Patients who have participated in another clinical trial within the last 3 months.
* Patients deemed unsuitable for participation in this clinical trial at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index(SPADI) Score | 6 months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The minimum value is 0 and the maximum value is 10. "0" means no pain and "10" means the worst pain imaginable in the pain section. "0" means no difficulty and "10" means so difficult it requires help in the pain section.

SECONDARY OUTCOMES:
Constant-Murley score | 6 months
  The Constant score assesses pain, function, ROM, and strength. Pain is allotted a maximum of 15 points, activities of daily living (function)20 points, ROM 40 points, and strength 25 points. The component scores are summated to achieve a maximum possible total score of 100.
Visual Analog Scale(VAS) pain in motion | 6 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 100mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Changes in the size of rotator cuff tears determined by MRI | 6 months
Changes in the size of rotator cuff tears determined by arthroscopy | 6 months
Adverse event | 6 months

OTHER OUTCOMES:
Change in degeneration score compared to baseline and the rate of change through histological examination | 6 months
  When tendon regeneration is identified in the lesion area through arthroscopic examination, a tissue sample approximately 2 mm in diameter is collected from the regenerated site and evaluated using the modified Astrom & Movin scoring system.
  The evaluation method consists of seven assessment variables(Fiber structure, Fiber arrangement, Rounding of the nuclei, Variations in cellularity, Increased vascularity, Decreased stainability, Hyalinization), each scored on a scale from 0 to 3, with 0 indicating normal and 3 representing the most severe abnormality. The scores are summed to calculate the tendon degeneration score, which ranges from 0 to 21. A score closer to 0 indicates normal tendon condition, while a score closer to 21 reflects severe degenerative changes.
STR (Short tandem repeat) analysis | 6 months
  STR analysis at post-injection
Visual Analog Scale_pain at night | 6 months
Visual Analog Scale(VAS) worst pain | 6 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 100mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Shoulder ROM (Forward flexion, Abduction, External rotation & Internal rotation at 0 degree) | 6 months
Muscle strength (lb) | 6 months
  The strength the supraspinatus, infraspinatus,and subscapularis was measured using a handheld electronic scale
Pulse rate (beats per minute) | 6 months
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using pulse rate
Blood Pressure (mmHg) | 6 months
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using blood pressure
CBC(complete blood count) | 6 months
  The measures are composite.
Usage amount of rescue medication | 6 months
  The total dosage of rescue medication administered to participants during the study period is measured to evaluate the amount of medication required to manage symptoms after treatment.
Frequency of rescue medication | 6 months
  The frequency of rescue medication usage is measured to assess how often participants required additional medication to manage symptoms during the study period.
Blood Glucose | 6 months
  Blood glucose levels are measured to assess glycemic control and detect hyperglycemia or hypoglycemia.
BUN/Creatinine Ratio | 6 months
  The ratio of blood urea nitrogen (BUN) to creatinine is measured to evaluate kidney function.
Serum Total Protein | 6 months
  Serum total protein levels are measured to evaluate overall protein status
Serum Albumin | 6 months
  Serum albumin levels are measured to assess liver function, nutritional status, and oncotic pressure regulation.
Serum total bilirubin | 6 months
  Serum total bilirubin levels are measured to evaluate liver function
Aspartate Transaminase/Alanine Transaminase(AST/ALT) | 6 months
  AST and ALT levels are measured to assess liver function
Serum Alkaline Phosphatase(ALP) | 6 months
  Serum ALP levels are measured to evaluate liver and bone health.
Serum Gamma-Glutamyl Transferase(γ-GTP) | 6 months
  Serum γ-GTP levels are measured to assess liver function
Serum creatine kinase(CK) | 6 months
  Serum creatine kinase levels are measured to assess muscle injury
Erythrocyte Sedimentation Rate(ESR) | 6 months
  ESR is measured to assess inflammation or detect inflammatory conditions
C-Reactive Protein(CRP) | 6 months
  Serum CRP levels are measured to evaluate acute inflammation
Urine pH Levels | 6 months
  Urine pH is measured to assess acidity or alkalinity of the urine. Lower values indicate increased acidity, while higher values indicate increased alkalinity. Normal range is typically 4.5-8.0.
Urine Specific Gravity | 6 months
  Urine specific gravity is measured to evaluate urine concentration or dilution. A value closer to 1.000 indicates more diluted urine, while higher values suggest more concentrated urine. protein
Urine Protein | 6 months
  Urine protein levels are measured to assess the presence of proteinuria. Normal range is typically negative or <20 mg/dL.
Urine Glucose | 6 months
  Urine glucose levels are measured to detect glycosuria. Normal range is negative.
Urine Bilirubin | 6 months
  Urine bilirubin levels are measured to assess liver function. Normal range is negative.
Urine Blood | 6 months
  Urine blood levels are measured to detect hematuria. Normal range is negative
Urine Ketone | 6 months
  Urine ketone levels are measured to detect ketonuria. Normal range is negative
Microscopic Analysis | 6 months
  Microscopic analysis of urine is performed to identify the presence of red blood cells (RBCs), white blood cells (WBCs), crystals, casts, or bacteria, which may indicate infection, inflammation, or other pathological conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, Korea, South Korea